CLINICAL TRIAL: NCT02989844
Title: Relapse Prophylaxis With IL-15 Super Agonist N-803 in Patients With Acute Myelogenous Leukemia and Myelodysplastic Syndrome Following Reduced Intensity Conditioning (RIC) Allogeneic Stem Cell Transplantation
Brief Title: Relapse Prophylaxis With N-803 for AML and MDS Pts Following Allo HSCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS058; MT2016-07 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2016-11-02; First posted 2016-12-12 (Estimated); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Acute Myelogenous Leukemia (AML); Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- N-803 (Experimental)
  Interventions: Drug: N-803

INTERVENTIONS:
Drug: N-803 — N-803 at 6 mcg/kg SQ Day 1 of a 4 week (28 day) cycle with ± 1 week window Continue N-803 every 4 weeks for 10 doses or until relapse, unacceptable toxicity, or patient refusal, whichever comes earlier.
  Other Names: Nant-803

SUMMARY:
This is a single-arm, multi-center Phase II trial using IL-15 super-agonist complex (N-803 formerly known as Alt-803) maintenance after allogeneic hematopoietic cell transplant (alloHCT) for acute myelogenous leukemia (AML) and myelodysplastic syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute myelogenous leukemia (AML) or myelodysplastic syndrome (MDS) for whom an allogeneic hematopoietic stem cell transplant using a reduced intensity conditioning is planned or has been performed and patient is prior to day 60 post-transplant.
2. Able to begin study treatment between day +42 and day +60 after the transplant and meets the following transplant related requirements:

   * Sustained neutrophil (ANC > 1000/mcL) and platelet (> 30,000/mcL) engraftment
   * >50% donor myeloid and lymphoid chimerism blood or bone marrow on most recent bone marrow (BM) evaluation
   * No evidence of recurrent disease on most recent bone marrow evaluation (day 21 or 28 post-transplant is acceptable)
   * No morphologic evidence of relapse (< 5% bone marrow blasts) on most recent BM evaluation (Day 21 or 28 post-transplant is acceptable)
   * Being followed in the outpatient setting (not an inpatient)
   * No plan of giving other anti-cancer treatment directed at diseases under study (i.e. maintenance therapy [e.g. sorafenib for FLT3m+ AML or hypomethylating therapy], additional therapy for MRD)
3. If acute GVHD is present it must be clinically improving on topical steroids and/or on low dose systemic steroids (≤ 0.3 mg/kg/day prednisone) and with clinical stability for at least 1 week prior to determination of eligibility. GVHD prophylaxis will be continued per individual institutional standard practice
4. One of the following donor graft sources used for the transplant:

   * Group 1: sibling donor
   * Group 2: haploidentical donor [with post-transplant cyclophosphamide]
   * Group 3: unrelated donor
   * Group 4: unrelated umbilical cord blood
5. Karnofsky performance status ≥ 70%
6. Adequate organ function within 14 days of study enrollment defined as:

   * Renal: serum creatinine: ≤ 2.0 mg/dL
   * Hepatic: SGOT ≤ 3 x upper limit of institutional normal (ULN)
7. Sexually active females of child-bearing potential and males with partners of child bearing potential must agree to use effective contraception during therapy and for 4 months after completion of therapy.
8. Voluntary written consent prior to the performance of any research related procedures

Exclusion Criteria:

1. Prior N-803 (previously known as ALT-803)
2. Pregnant or breastfeeding - N-803 is an investigational agent. Women of child bearing potential must have a negative pregnancy test at screening.
3. Class II or greater New York Heart Association Functional Classification criteria or serious cardiac arrhythmias likely to increase the risk of cardiac complications of cytokine therapy (e.g. ventricular tachycardia, frequent ventricular ectopy, or supraventricular tachyarrhythmia requiring chronic therapy)
4. Marked baseline prolongation of QT/QTc interval (e.g. demonstration of a QTc interval > 500 milliseconds)
5. Active uncontrolled bacterial, fungal, or viral infections - all prior infections must have resolved following optimal therapy and must be afebrile for at least 24 hours at time of enrollment.
6. Active autoimmune disease requiring immunosuppressive therapy (GVHD prophylaxis is permitted per institutional practice)
7. History of severe asthma and currently on chronic medications (mild asthma requiring inhaled steroids only is eligible)
8. Received any investigational agent within the 14 days before the start of study treatment (1st dose of N-803)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2022-03-19 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Brunstein, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-803
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | N-803
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Relapse
Description: Efficacy of N-803 as measured by the cumulative incidence of relapse between the 1st dose of N-803 and 2 years after a reduced intensity conditioning (RIC) allogeneic hematopoietic cell transplant (alloHCT)
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | N-803
Number analyzed (Participants) | 20
Percentage of participants | 30 [12 to 51]

2. Secondary Outcome: Incidence of Adverse Events
Description: Frequency of all adverse
Time Frame: 12 months
Measure: Number; unit: Count of events
Arm/Group | N-803
Number analyzed (Participants) | 20
Count of events | 567

3. Secondary Outcome: Incidence of Acute Graft-versus-host Disease
Description: Incidence of grade 2-4 and grade 3-4 acute graft-versus-host-disease (GVHD)
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | N-803
Number analyzed (Participants) | 20
Percentage of participants
  Grade 2-4 GVHD | 10 [2 to 28]
  Grade 3-4 GVHD | 0 [0 to 100]

4. Secondary Outcome: Incidence of Acute Graft-versus-host Disease
Description: Incidence of grade 2-4 and grade 3-4 acute graft-versus-host-disease (GVHD)
Time Frame: Day 180
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | N-803
Number analyzed (Participants) | 20
Percentage of participants
  Grade 2-4 GVHD | 15 [4 to 34]
  Grade 3-4 GVHD | 5 [0 to 21]

5. Secondary Outcome: Chronic GVHD
Description: Incidence of acute graft-versus-host disease
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | N-803
Number analyzed (Participants) | 20
Percentage of participants | 15 [4 to 34]

6. Secondary Outcome: Minimal Residual Disease (MRD)
Description: Incidence of minimal residual disease (MRD) post-transplant
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | N-803
Number analyzed (Participants) | 20
Percentage of participants | 26 [12 to 49]

7. Secondary Outcome: Overall Survival
Description: Incidence of overall survival at one year
Time Frame: 1 year post transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | N-803
Number analyzed (Participants) | 20
Percentage of participants | 85 [71 to 99]

8. Secondary Outcome: Non-Relapse Mortality
Description: Incidence of non-relapse mortality
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | N-803
Number analyzed (Participants) | 20
Percentage of participants | 5 [0 to 21]

9. Secondary Outcome: Relapse
Description: Incidence of relapse at 2 years after alloHCT stratified by number of doses of N-803 (1-3 or 4-10)
Time Frame: 2 Years
Population: Intent is to compare the percentage of participants with relapse stratified according the number of doses of N-803 that were administered.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | N-803
Number analyzed (Participants) | 20
Percentage of participants
  1-3 doses of N-803: number analyzed (Participants) | 8
  1-3 doses of N-803 | 62 [18 to 88]
  4-10 doses of N-803: number analyzed (Participants) | 12
  4-10 doses of N-803 | 17 [2 to 43]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | N-803
All-Cause Mortality (participants affected / at risk) | 3/20
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-803 (N=20)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Infections and infestations - Other, (Infections and infestations) | 1 (1)
Immune system disorders - Other, (Immune system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-803 (N=20)
Anemia (Blood and lymphatic system disorders) | 20 (22)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 4 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 17 (17)
Edema limbs (General disorders) | 8 (8)
Fatigue (General disorders) | 12 (12)
Fever (General disorders) | 8 (8)
Injection site reaction (General disorders) | 20 (47)
Gait disturbance (General disorders) | 4 (4)
Injection site reaction (General disorders) | 20 (48)
Pain (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2)
Allergic reaction (Immune system disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3)
Lung infection (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 7 (7)
Vulval infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Alanine aminotransferase increased (Investigations) | 5 (5)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 10 (10)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 8 (8)
Lymphocyte count decreased (Investigations) | 5 (5)
Neutrophil count decreased (Investigations) | 20 (21)
Platelet count decreased (Investigations) | 20 (46)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 20 (39)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (15)
Hypermagnesemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 9 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (10)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 8 (8)
Hypertension (Vascular disorders) | 20 (76)
Hypotension (Vascular disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT02989844/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT02989844/ICF_001.pdf